CLINICAL TRIAL: NCT00391144
Title: Intravitreal Avastin Injection for the Treatment of Choroidal Neovascularization Secondary to Pattern Dystrophy
Brief Title: Avastin for CNV Secondary to Pattern Dystrophy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Trieste (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1/2006
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Last update posted 2006-10-23 (Estimated); Status verified 2006-10

CONDITIONS: Choroidal Neovascularization Secondary to Pattern Dystrophy
Keywords: Pattern Dystrophy; Choroidal Neovascularization; Intravitreal Avastin Injection
MeSH Terms: conditions — Choroidal Neovascularization

INTERVENTIONS:
Procedure: intravitreal triamcinolone injection of avastin (1.25 mg)

SUMMARY:
The natural history of subfoveal CNV secondary to Pattern Dystrophy is little understood, but it seems that visual function may be preserved only in the short-term follow-up, with progressive deterioration thereafter.

Photodynamic therapy with verteporfin is the most studied therapeuthic option for this kindf of lesion, but unfortunately, this approach does not appear to guarantee long-term vision stabilization, and alternative therapies should be investigated.

DETAILED DESCRIPTION:
Diagnosis of Pattern Dystrophy Diagnosis of subfoveal CNV Intravitreal injection of avastin (1.25 mg) in operating room under sterile condition.

Retreatment on the basis of the detection of disease progression and of lack of central retinal thickness reduction on OCT.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of RPD (hyperpigmented yellowish-greyish network, other family members sharing RPD, normal electroretinogram and normal/subnormal electrooculogram)
* classic or occult CNV involving the foveal avascular zone's geometric centre

Exclusion Criteria:

* conditions other than RPD
* intraocular surgery or capsulotomy within the last 2 or 1 months
* pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5
Dates: Start 2006-07; Study Completion 2006-10

PRIMARY OUTCOMES:
number of eyes with <15 letter loss (approximately <3 lines) at 6-month examination compared with the baseline value
numeber of eyes with <15 letter loss at 12-month examinations, compared with the baseline value.

SECONDARY OUTCOMES:
CNV progression
number of injections.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio B Parodi, MD, Principal Investigator — Clinica Oculistica, Azienda Ospedaliero-Universitaria di Trieste; Pierluigi Iacono, MD, Principal Investigator — Clinica Oculistica, Azienda Ospedaliero-Universitaria di Trieste; Giuseppe Ravalico, MD, Study Director — Clinica Oculistica, Azienda Ospedaliero-Universitaria di Trieste
Locations (1):
- Clinica Oculistica, Azienda Ospedaliero-Universitaria di Trieste, Trieste, TS, Italy

REFERENCES:
- [Result] Parodi MB, Liberali T, Pedio M, Francis PJ, Piccolino FC, Fiotti N, Romano M, Ravalico G. Photodynamic therapy of subfoveal choroidal neovascularization secondary to reticular pattern dystrophy: three-year results of an uncontrolled, prospective case series. Am J Ophthalmol. 2006 Jun;141(6):1152-4. doi: 10.1016/j.ajo.2006.01.038. PMID 16765697
- [Result] Da Pozzo S, Parodi MB, Toto L, Ravalico G. Occult choroidal neovascularization in adult-onset foveomacular vitelliform dystrophy. Ophthalmologica. 2001 Nov-Dec;215(6):412-4. doi: 10.1159/000050899. PMID 11741106
- [Result] Battaglia Parodi M, Da Pozzo S, Ravalico G. Photodynamic therapy for choroidal neovascularization associated with pattern dystrophy. Retina. 2003 Apr;23(2):171-6. doi: 10.1097/00006982-200304000-00006. PMID 12707595
- [Result] Battaglia Parodi M, Di Crecchio L, Ravalico G. Vascularized pigment epithelial detachment in adult-onset foveomacular vitelliform dystrophy. Eur J Ophthalmol. 2000 Jul-Sep;10(3):266-9. doi: 10.1177/112067210001000315. PMID 11071039
- [Result] Battaglia Parodi M, Iustulin D, Russo D, Ravalico G. Adult-onset foveomacular vitelliform dystrophy and indocyanine green videoangiography. Graefes Arch Clin Exp Ophthalmol. 1996 Mar;234(3):208-11. doi: 10.1007/BF00462035. PMID 8720722
- [Derived] Parodi MB, Iacono P, Cascavilla M, Zucchiatti I, Kontadakis DS, Bandello F. Intravitreal bevacizumab for subfoveal choroidal neovascularization associated with pattern dystrophy. Invest Ophthalmol Vis Sci. 2010 Sep;51(9):4358-61. doi: 10.1167/iovs.10-5237. Epub 2010 Apr 7. PMID 20375343